CLINICAL TRIAL: NCT00214812
Title: An Imaging Trial of the Distribution of Topical Gel in the Human Vagina: Assessment of Bare Spots
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosyn (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RRU-005
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: HEC placebo gel

SUMMARY:
This study will assess the distribution of a microbicidal gel in the vagina and confirm the presence of bare spots. MRIs will be done with and without the addition of the MRI contrast Gadolinium to the microbicide in order to determine whether the bare spots are an artifact of the MRI technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 -45 year old women
* normal Pap smear
* not pregnant

Exclusion Criteria:

* abnormal pelvic exam
* history of claustrophobia
* allergy to product formulation
* pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2005-06

PRIMARY OUTCOMES:
Presence or absence of bare spots with and without Gd.
Quantification and location of bare spots.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Barnhart, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Reproductive Research Unit, U of Penn Medical Center, Philadelphia, Pennsylvania, United States